CLINICAL TRIAL: NCT05301075
Title: Rhomboid Intercostal and Subserratus Plane (RISS) Block on Postoperative Painafter Open Nephrectomy Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: N-74-2021
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Rhomboid Intercostal Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator): patients will receive sham block.
  Interventions: Drug: Rhomboid Intercostal and Sub-Serratus block
- RISS group (Active Comparator): will receive Rhomboid Intercostal and Sub-Serratus block under ultrasound guidance
  Interventions: Drug: Rhomboid Intercostal and Sub-Serratus block

INTERVENTIONS:
Drug: Rhomboid Intercostal and Sub-Serratus block — Rhomboid Intercostal and Sub-Serratus block under ultrasound guidance

SUMMARY:
Rhomboid intercostal block (RIB) is a new interfascial plane block describe by Elsharkawy et al. in 2016. The region described is understood because the triangle of auscultation that's bounded medially by inferior a part of the trapezius, inferiorly by the superior border of latissimus dorsi, and laterally by the medial border of the scapula. In this ultrasound-guided block, the local anaesthetic drug is run between the rhomboid major and therefore the intercostal fascia at the extent of T6-T7 and provides analgesia of T3-T8 dermatomes

ELIGIBILITY:
* Inclusion criteria Adult patients between 18-60 years. Genders eligible for study: both sexes ASA physical status I and II Undergoing open nephrectomy surgery
* Exclusion criteria Patient refusal Contraindications to regional anesthesia Known allergy to local anesthetics Bleeding disorders Use of any anti-coagulants Inability to provide informed consent ASA III-IV

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-21 (Estimated); Primary Completion 2023-08-13 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
nalbuphine consumption i | 24 hours
  Postoperative nalbuphine consumption

SECONDARY OUTCOMES:
nalbuphine consumption. | 2 hours
  intraoperative nalbuphine consumption.
Patient's satisfaction | 24 hours
  using 1-4 scales (1, bad; 2, moderate; 3, good; 4, excellent;

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
still working